CLINICAL TRIAL: NCT04507061
Title: A Randomized, Double-blind, Placebo-controlled, Multi-center Study to Assess the Safety and Efficacy of Individually Titrated Oral Doses of Runcaciguat in Subjects With Clinical Diagnosis of Chronic Kidney Disease With Diabetes and/or Hypertension and at Least One Cardiovascular Comorbidity
Brief Title: Study on the Safety of the Drug Runcaciguat and How Well it Works When Given at the Highest Dose as Tolerated by Individual Patient Whose Kidneys Are Not Working Properly and Suffering at the Same Time From High Blood Sugar and/or High Blood Pressure and a Disease of the Heart and the Blood Vessels.
Acronym: CONCORD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 18748; 2019-003297-53 (EudraCT Number)
Record Dates: First submitted 2020-08-06; First posted 2020-08-10 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — BAY 1101042

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- runcaciguat (Experimental): Participant randomized to this arm will be up-titrated. A 30-day safety follow up will be performed after end of treatment or after early discontinuation from the study.
  Interventions: Drug: runcaciguat
- Placebo (Placebo Comparator): Participant randomized to this arm will be sham-titrated. A 30-day safety follow up will be performed after end of treatment or after early discontinuation from the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: runcaciguat — Titrated dose of active dose 1, dose 2, dose 3, dose 4 of runcaciguat will be administered orally once a day.
  Arms: runcaciguat
Other: Placebo — Sham-titrated dose of matching placebo will be administered orally once a day.
  Arms: Placebo

SUMMARY:
Researchers in this study want to learn more about the safety of the drug runcaciguat and how well it works when given at the highest dose as tolerated by the individual patient whose kidneys are not working properly and suffering at the same time from high blood sugar and/or high blood pressure and a disease of the heart and the blood vessels. Runcaciguat is a new drug under development for the improvement of kidney function. It works by activating proteins that helps to dilate blood vessels, including vessels in the kidneys. This can improve blood flow in kidney and may slow down the progression of kidney disease. This dilative effect can also influence the heart rate and blood pressure. Researchers also wants to find the best dose of the drug during the study.

Participants in this study will receive either runcaciguat or placebo tablets every morning for 8 weeks. A placebo looks like the study drug but does not have any active medicine in it. On a weekly basis, the dose of the runcaciguat will be increased step by step. In total, participants will visit the doctors about 10 times, and the observation will last for about 16 weeks. Blood and urine samples will collected from the participants.

ELIGIBILITY:
Inclusion Criteria:

Age - Participant must be ≥ 45 of age inclusive, at the time of signing the informed consent.

Type of Participant and Disease Characteristics

- Participants who have:

* history of any of the following:

  * type 2 diabetes mellitus as defined by the American Diabetes Association (on treatment with glucose-lowering medications and/or insulin) for at least 2 years, and/or;
  * diagnosis of hypertension (defined as systolic blood pressure [BP] values ≥ 140 mmHg and/or diastolic BP values ≥90 mmHg) and on hypertension medication for at least 5 years;
* established atherosclerotic cardiovascular disease (e.g. coronary artery disease, peripheral arterial disease, cerebrovascular disease) or heart failure;
* a clinical diagnosis of chronic kidney disease (CKD) based on all of the following criteria:

  * (estimated) glomerular filtration rate (eGFR) ≥ 25 mL/min/1.73 m^2 but ≤ 60 mL/min/1.73 m^2 (acc. Percentage of decrease in eGFR [CKD EPI]);
  * persistent high albuminuria defined as urine albumin-to-creatinine ratio [UACR] of between 30 mg/g and 3000 mg/g in 2 first morning void samples (collected at least 1 week apart);
  * Stable treatment with angiotensin-converting enzyme inhibitor (ACEi) or angiotensin-receptor blocker (ARB) for the participant maximum tolerated labelled daily dose and otherwise stable antihypertensive treatment both for at least 3 months before randomization, without any adjustments to this therapy for at least 4 weeks prior to randomization;
* Diabetes patients that are on SGLT2-inhibitor (SGLT: sodium glucose transport protein) have to be on stable treatment for at least 3 months before Screening visit.

Exclusion Criteria:

* Known non-diabetic and non-hypertension related renal diseases as autosomal dominant polycystic kidney disease, bilateral clinically relevant renal artery stenosis, lupus nephritis, or ANCA-associated vasculitis, IgA nephropathy without hypertension, or any other secondary glomerulonephritis;
* Clinical diagnoses of heart failure and persistent symptoms (New York Heart Association (NYHA class III - IV);
* Uncontrolled hypertension indicated by >160 mmHg systolic BP or ≥ 100 mmHg diastolic BP;
* History of secondary hypertension (i.e., renal artery stenosis, primary aldosteronism, or pheochromocytoma);
* Stroke, transient ischemic cerebral attack, acute coronary syndrome, or hospitalization for worsening heart failure, in the last 3 months prior to the planned randomization;
* Dialysis for acute renal failure within the previous 6 months prior to the planned randomization;
* Renal allograft in place or a scheduled kidney transplant within the next 18 weeks (being on a waiting list does not exclude the subject);
* Hepatic insufficiency classified as Child-Pugh B or C or other significant liver disease (e.g., acute hepatitis, chronic active hepatitis, cirrhosis as indicated by e.g. aspartate aminotransferase [AST] or Alanine aminotransferase [ALT] >3x upper limit of norm [ULN]);
* Active malignancy other than treated squamous cell, carcinoma in situ, or basal cell carcinoma of the skin Prior/Concomitant Therapy;
* Any surgical or medical condition, which in the opinion of the investigator, may place the patient at higher risk from his/her participation in the study, or is likely to prevent the patient from complying with the requirements of the study or completing the study including but not limited to:

  1. History of active inflammatory bowel disease within the last 6 months before randomization;
  2. Major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection;
  3. Gastro-intestinal ulcers and/or gastrointestinal or rectal bleeding within last 6 months before randomization;
  4. Pancreatic injury or pancreatitis within the last 6 months before randomization;
* Non diabetic patients treated with SGLT-2 (SGLT:sodium glucose transport protein) inhibitors;
* Combination use of ACEi and ARB within 3 months prior to randomization;
* Concomitant therapy with nitrates, PDE5 inhibitors including nonspecific inhibitors (e.g. dipyridamole and theophylline), soluble guanylate cyclase [sGC] stimulators, renin inhibitors (within 4 weeks prior to randomization);
* Participation in another clinical study or treatment with another investigational product 90 days prior to randomization;
* Previous randomization in this study;
* hemoglobin A1c (HbA1c) >11%;

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2022-04-05 (Actual)

PRIMARY OUTCOMES:
Mean change in urinary albumin-to-creatinine ratio (UACR) from baseline to the average of multiple time points during treatment | From baseline up to day 57 (± 3)

SECONDARY OUTCOMES:
Number of subjects with treatment emergent adverse event (TEAE) | From first treatment administration up to end of follow up (Day 87±7)
Number of subjects with early discontinuations | From first treatment administration up to end of treatment (Day 57±3)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (70):
- Austria (5):
  - Medizinische Universität Innsbruck, Innsbruck
  - Klinik Landstraße - Krankenhaus Rudolfstiftung, Vienna
  - Zentrum f. klinische Studien Dr. Hanusch GmbH, Vienna
  - Universitätsklinikum AKH Wien, Vienna
  - Klinik Hietzing, Vienna
- Belgium (4):
  - OL Vrouwziekenhuis - Campus Aalst, Aalst
  - Hôpital Erasme/Erasmus Ziekenhuis, Bruxelles - Brussel
  - UZ Gent, Ghent
  - UZ Leuven Gasthuisberg, Leuven
- Bulgaria (7):
  - Med Centre Diamedical 2013, Dimitrovgrad
  - Multiprofile Hospital for Active Treatment Medline Clinic, Plovdiv
  - MHAT Sveta Karidad, Plovdiv
  - MHAT Dr. Bratan Shukerov AD, Smolyan
  - MHAT "Knyaginya Klementina - Sofia"EAD, Sofia
  - MC Kalimat, Sofia
  - MCOMH Preventsia-2000, Stara Zagora
- Denmark (6):
  - Region Nordjylland | Aalborg University Hospital - Cardiology Department, Aalborg
  - Steno Diabetes Center Copenhagen, Herlev
  - Regionshospitalet Gødstrup, Herning
  - Holbæk Sygehus, Holbæk
  - Sygehus Lillebaelt | Kolding Sygehus - Medicinske Sygdomme, Kolding
  - Odense Universitetshospital, Endokrinologisk Afd. M, Odense C
- Finland (5):
  - StudyCor Oy, Jyväskylä
  - Diagnos Klaukkalan Lääkäriasema, Klaukkala
  - Satucon / Kuopion Työterveys, Kuopio
  - Omena Terveys Oy, Seinäjoki
  - Turun yliopistollinen keskussairaala, Turku
- Germany (5):
  - Klinikum der Universität Würzburg, Würzburg, Bavaria
  - Herz- und Diabeteszentrum Nordrhein-Westfalen (HDZ NRW), Bad Oeynhausen, North Rhine-Westphalia
  - DaVita Clinical Research Deutschland GmbH, Düsseldorf, North Rhine-Westphalia
  - InnoDiab Forschung GmbH, Essen, North Rhine-Westphalia
  - Medamed Studienambulanz GmbH, Leipzig, Saxony
- Israel (8):
  - Barzilai Medical Center | Nephrology & Hypertension Dept., Ashkelon
  - Lady Davis Carmel Medical Center, Haifa
  - Edith Wolfson Medical Center, Holon
  - Hadassah Hebrew University Hospital Ein Kerem, Jerusalem
  - Health Corporation of Galilee Medical Center, Nahariya
  - Clalit Health Services Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Poriya Medical Center | Nephrology and Hypertension Dept., Tiberius
- Italy (6):
  - A.O.U. Luigi Vanvitelli, Napoli, Campania
  - A.O.U. di Bologna Policlinico S.Orsola Malpighi, Bologna, Emilia-Romagna
  - IRCCS Ospedale Policlinico San Martino, Genoa, Liguria
  - Istituto Ricerche Farmacologiche Mario Negri IRCCS, Bergamo, Lombardy
  - Ospedale San Raffaele s.r.l., Milan, Lombardy
  - IRCCS Centro Cardiologico Monzino S.p.A, Milan, Lombardy
- Centralny Szpital Kliniczny MSWiA w Warszawie, Warsaw, Poland
- Slovakia (3):
  - FMC-dialyzacne sluzby, s.r.o. - Kosice, Košice
  - BIODIAL, spol. s r.o., Púchov
  - Medivasa s.r.o., Žilina
- Spain (8):
  - Complejo Hospitalario Universitario de Ferrol | Hospital Naval - Unidad de Hipertensión Arterial, Ferrol, A Coruña
  - Complejo Hosp. Univ. A Coruña | Endocrinologia y Nutricion, A Coruña
  - Hospital del Mar, Barcelona
  - Ciutat Sanitaria i Universitaria de la Vall d'Hebron, Barcelona
  - Hospital Quirón, Barcelona
  - Hospital Universitario Virgen de las Nieves|Medicina Interna, Granada
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
- Sweden (4):
  - PTC-Primary care Trial Center, Gothenburg
  - Clemenstorget Hjärtmottagning, Lund
  - Akademiska Sjukhuset Njurmottagningen, Uppsala
  - ClinSmart, Uppsala
- Ukraine (8):
  - Medical center LLC " Fresenius medical care Ukraine", Cherkasy
  - Dnepropetrovsk regional hospital n.a. I. I. Mechnikov, Dnipro
  - Private enterprise private production company " Acinus", Kropyvnytskyi
  - Kyiv City Center of Nephrology and Dialysis, Kyiv
  - Medical Center of Edelweiss Medics LLC, Kyiv
  - Volyn Regional Clinical Hospital, Lutsk
  - Ternopil Regional Clinical Hospital, Ternopil
  - Zaporizhzhia Regional Clinical Hospital, Zaporizhzhya

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access.
  As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Derived] Gansevoort RT, Wheeler DC, Deben FM, Speeckaert M, Thomas D, Berger M, Klein S, Friedrichs F, Paraschin K, Schmieder RE. The soluble guanylate cyclase activator runcaciguat significantly improves albuminuria in patients with chronic kidney disease: a randomized placebo-controlled clinical trial. Nephrol Dial Transplant. 2025 May 30;40(6):1147-1160. doi: 10.1093/ndt/gfae261. PMID 39656628
- [Derived] Kraehling JR, Benardeau A, Schomber T, Popp L, Vienenkoetter J, Ellinger-Ziegelbauer H, Pavkovic M, Hartmann E, Siudak K, Freyberger A, Hagelschuer I, Mathar I, Hueser J, Hahn MG, Geiss V, Eitner F, Sandner P. The sGC Activator Runcaciguat Has Kidney Protective Effects and Prevents a Decline of Kidney Function in ZSF1 Rats. Int J Mol Sci. 2023 Aug 25;24(17):13226. doi: 10.3390/ijms241713226. PMID 37686032
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/